CLINICAL TRIAL: NCT00169689
Title: Therapeutic and Biological Effects of High Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) in Schizophrenia
Brief Title: Repetitive Transcranial Magnetic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Cordes, Joachim, Heinrich-Heine University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS_S_01; TMS_01
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Schizophrenia
Keywords: schizophrenia, rTMS
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- rTMS (Sham Comparator): sham coil system versus verum rTMS stimulation
  Interventions: Procedure: rTMS, "repetitive transcranial magnetic stimulation"; Other: rTMS

INTERVENTIONS:
Procedure: rTMS, "repetitive transcranial magnetic stimulation" — 10 Hz rTMS (10.000 stimuli) over left dorsolateral prefrontal cortex
Other: rTMS — repetitive transcranial magnetic stimulation, 10 Hz, 10.000 stimuli, 2 weeks

SUMMARY:
The study is a prospective, randomized, double-blind sham-controlled study.

DETAILED DESCRIPTION:
The principal objective of this trial is to investigate the effect of left prefrontal high frequency rTMS on negative symptoms in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for schizophrenia
* age between 18 and 60
* informed consent
* right handed patient
* no change of antipsychotic treatment > 2 weeks before recruitment

Exclusion Criteria:

* seizures, epilepsy
* history of severe head injury
* status post implantation of a cardiac pacemaker or other electronic devi-ses

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2003-06; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression; | November 2007

SECONDARY OUTCOMES:
Global psychosocial functioning (GAF), PANSS-Negative Subscale,changes in EEG, heart rate variability, cortisol daytime profile, catecholamines, cognitive functioning | November 2007

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Cordes, MD, Principal Investigator — Department of Psychiatry and Psychotherapy at the Heinrich-Heine-University Düsseldorf,Rhineland State Clinics Düsseldorf, Bergische Landstraße 2, 40629 Düsseldorf, Germany; PD Dr. W Wölwer, Principal Investigator — Heinrich-Heine-University; PD Dr. MW Agelink, Principal Investigator — Department of Psychiatry Herford
Locations (1):
- Joachim Cordes, Düsseldorf, Rhineland, Germany

REFERENCES:
- [Result] Cordes J, Arends M, Mobascher A, Jänner M, Wölwer W, Krieger K, Agelink MW, Klimke A, Brinkmeyer J. Left prefrontal high frequency repetitive transcra-nial magnetic stimulation (rTMS) and the effect on schizophrenic psychopathol-ogy. European Archives of Psychiatry and Clinical Neuroscience 2004; Vol. 254, Suppl. 1: 11. Cordes J, Brinkmeyer J, Kotrotsios G, Arends M, Mobascher A, Agelink MW, Wölwer W. The effect of high frequency repetitive transcranial magnetic stimula-tion (rTMS) on negative symptoms and electrophysiological correlates of facial affect recognition in schizophrenia. Schizophrenia Bulletin 2005 b; 31 (2): 510.
- [Derived] Wolwer W, Lowe A, Brinkmeyer J, Streit M, Habakuck M, Agelink MW, Mobascher A, Gaebel W, Cordes J. Repetitive transcranial magnetic stimulation (rTMS) improves facial affect recognition in schizophrenia. Brain Stimul. 2014 Jul-Aug;7(4):559-63. doi: 10.1016/j.brs.2014.04.011. Epub 2014 May 9. PMID 24857264
- [Derived] Cordes J, Thunker J, Agelink MW, Arends M, Mobascher A, Wobrock T, Schneider-Axmann T, Brinkmeyer J, Mittrach M, Regenbrecht G, Wolwer W, Winterer G, Gaebel W. Effects of 10 Hz repetitive transcranial magnetic stimulation (rTMS) on clinical global impression in chronic schizophrenia. Psychiatry Res. 2010 May 15;177(1-2):32-6. doi: 10.1016/j.psychres.2009.01.014. Epub 2010 Apr 8. PMID 20378181